CLINICAL TRIAL: NCT03841344
Title: A Prospective Study Comparing the REpeatability and Sensitivity to Change of Non-invasive Endpoints in Pulmonary arterIal hypeRtEnsion
Brief Title: Repeatability and Sensitivity to Change of Non-invasive Endpoints in PAH
Acronym: RESPIRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Andy J Swift, Wellcome Trust Clincial Research Career Development Fellow - principle investigator, University of Sheffield
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STH18285
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Walk Test

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers (Active Comparator): MRI 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP
  Interventions: Device: MRI
- Treatment naive patients (Active Comparator): MRI 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP
  Patients diagnosed with PAH initiating PAH therapy for the first time
  Interventions: Device: MRI
- Treatment change patients (Active Comparator): MRI 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP
  Patients diagnosed with PAH, currently on PAH therapy who are undergoing an escalation of PAH therapy
  Interventions: Device: MRI
- Stable patients (Active Comparator): MRI 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP
  Patients with PAH who are NOT undergoing changes in their treatment regime
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Evaluation of the utility of candidate endpoints in PAH trials
  Other Names: 6 minute walk test, incremental shuttle walk test, NT-ProBNP and BNP

SUMMARY:
Pulmonary arterial hypertension (PAH) is progressive life limiting disease with a median survival of less than 3 years without treatment. Current drug trials in PAH commonly use simple tests for example the 6-minute walk test, blood tests such as N-terminal pro-brain-type natriuretic peptide (NT-pro-BNP) and BNP, and haemodynamic measures such as PAP and PVR obtained by RHC as endpoints. These tests are surrogate markers of disease severity in patients with pulmonary hypertension. There is now evidence suggesting that magnetic resonance imaging (MRI) may be helpful in the follow up of patients with PAH with high accuracy for the detection of treatment failure, this is because MRI can track changes occurring in the heart by direct visualisation of cardiopulmonary morphology and function, an advantage over existing methods. However, the reproducible of MRI measurements in patients with PAH is not known, and the comparative repeatability of MRI in relation to traditional candidate endpoints such as walk tests and blood tests used in drug trials is not known.

DETAILED DESCRIPTION:
Background:

Pulmonary arterial hypertension (PAH) is a rare but severe and progressive disorder, with a prevalence of approximately 50 in 1,000,000 of the population. The condition is incurable with high morbidity and mortality despite the development of effective treatment options. The emergence of goal orientated therapy initially focused interest on prognostic markers that can both inform the clinician regarding disease severity at presentation and be used to follow-up response to therapy and aid in decisions regarding listing for transplantation. A number of effective therapies are available but are very expensive and there is an urgent need for non-invasive and specific markers to assess treatment response and guide therapy. Accurate follow up with reproducible measurements of the heart and pulmonary vasculature are essential in order to accurately characterise treatment response.

Magnetic resonance imaging (MRI) a non-ionising and non-invasive technique provides accurate and reproducible information on cardiac morphology and function. MR imaging is becoming an established technique in the evaluation of patients with PAH, allowing direct visualisation and accurate analysis of the structure and function of the right ventricle (RV). There is a pressing need to validate and standardise MRI methods in pulmonary hypertension to allow clinical translation nationally and internationally and to support trials of novel disease modifying therapies.

Aims:

The aim of this study is to determine the repeatability and capability of detecting change of MR imaging measurements in comparison with walk tests and blood tests in patients with PAH, and define the optimal MRI analysis protocol for use in clinical practice and in future studies in PAH.

Objectives:

* Determine the inter-observer and inter-scan variability of MRI in healthy volunteers and patients with PAH
* Compare the inter-observer and inter-scan variability of MRI with walk tests and blood tests, in healthy volunteers and patients with PAH
* Determine the capability of MRI to detect change in PAH patients with start or change of therapy in comparison to walk test and blood test data.
* Compare MRI endpoints with associated clinical data including haemodynamic measures obtained by right heart catheterisation

Plan of investigation:

Participants:

Participants from the following groups will be recruited:

* Treatment naïve patients with PAH
* Patients with PAH undergoing changes in their treatment regime
* Patients with PAH who are NOT undergoing changes in their treatment regime
* Healthy volunteers will be recruited.

PAH treatment will be as per standard of care. No new therapies are being tested.

Sample sizes:

Recruit sufficient incident treatment naïve patients with PAH and patients with PAH on monotherapy whose treatment is to be changed to achieve approximately 40 completers. This number is based on prior MRI reproducibility studies investigating the reproducibility of right ventricular measurements in healthy subjects and in those with cardiovascular disease. It is planned that at least 30% of patients will be treatment naïve. 20 healthy volunteer subjects will be recrited

Visit schedule Patients with pulmonary arterial hypertension Baseline study visit: During the baseline visit, blood draw, 6 minute walk test (+/- shuttle walk test) and cardiopulmonary MRI will be performed.

Follow-up visit: A follow-up visit will then occur at any time between 1 and 12 months after baseline. Patients with PAH, will be admitted for a one or two day visit. Cardiopulmonary MRI, blood draw, 6 minute walk test (+/- shuttle walk test) in the morning. Patients will take their usual medications approximately 1 hour prior to their MRI. These investigations will be repeated in the afternoon in the same way and in the same order. Patients will refrain from, exercise, caffeinated drinks and alcohol, between investigations.

Healthy volunteers Recruited by open advertisement within the hospital and university. Male or female subjects aged 18-60 years. Subjects will attend for a half day baseline visit for MRI, walk tests and blood tests. The follow up visit, including MRI, blood draw and walk test(s) will be as described for patients with PAH.

End points:

The MRI protocol will include measurement of candidate markers from the right heart and pulmonary vasculature:

I. Biventricular volume, mass and function. Analysis from both the 4 chamber and short axis images. Analyses will include and exclude trabecular mass.

II. Interventricular septal curvature and left ventricular eccentricity III. Pulmonary arterial flow, pulmonary arterial area change and pulsatility IV. Dynamic contrast enhanced perfusion imaging (first pass pulmonary transit time, full-width-half-maximum, delayed enhancement washout time) V. Myocardial and pulmonary tissue characteristics pre and post contrast T1 mapping of heart and lungs and myocardial late gadolinium enhancement pattern VI. Other MRI endpoints including composite measures

Analysis of MRI will be undertaken blinded to the patient's covariate data (walk tests and blood tests). Two experienced (one primary, one secondary) independent observers will analyse all the MRI studies. In the event of discrepancy between observers, the images will be reviewed by a third observer (radiologist) and all three observers should reach consensus.

Biomarker and walk test evaluation - The patient will be bled via a needle or cannula. Whenever possible, blood tests will precede the walk test and MRI. Candidate prognostic biomarkers, Pro NT BNP and BNP, will be tested. Incremental shuttle walk test and the 6 minute walk test will be performed >45 minutes apart and both tests will be repeated in the afternoon to determine the between measurement reproducibility for comparison with MRI. Walk tests will be performed in accordance with standard protocols.

ELIGIBILITY:
Patients with PAH

Inclusion Criteria:

* PAH subject is diagnosed with Group 1 pulmonary arterial hypertension, including IPAH, hereditable and CTD, and PAH associated with portal hypertension
* Mean pulmonary arterial pressure ≥ 25 mmHg
* Pulmonary arterial wedge pressure ≤ 15 mmHg

Exclusion Criteria:

* Inability to perform the study protocol
* Significant comorbidity where in the opinion of the clinician this is a significant contributor to the patients PAH
* Pregnancy
* Allergy to contrast medium
* Contraindication to MRI (as per standard screening questionnaire)
* Significant lung disease.
* Known Hep B,C, HIV

Healthy volunteers

Inclusion criteria:

* Male or female aged between 18 years and 60 years
* Currently healthy as determined by a responsible physician
* No significant history of lung or cardiac disease and normal BNP.
* Capable of giving written informed consent.
* Subject is >50kg with a body mass index within the range 18.0 to 32kg/m2.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2019-05-20 (Estimated)

PRIMARY OUTCOMES:
Repeatability of endpoints | Measurements repeated within 24 hours
  Repeatability of MRI, 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP
Sensitivity to change of endpoints | Follow up visits performed at 1-12 months
  Sensitivity to change of MRI, 6 minute walk test, incremental shuttle walk test, NT-Pro BNP and BNP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alabed S, Alandejani F, Dwivedi K, Karunasaagarar K, Sharkey M, Garg P, de Koning PJH, Toth A, Shahin Y, Johns C, Mamalakis M, Stott S, Capener D, Wood S, Metherall P, Rothman AMK, Condliffe R, Hamilton N, Wild JM, O'Regan DP, Lu H, Kiely DG, van der Geest RJ, Swift AJ. Validation of Artificial Intelligence Cardiac MRI Measurements: Relationship to Heart Catheterization and Mortality Prediction. Radiology. 2022 Oct;305(1):68-79. doi: 10.1148/radiol.212929. Epub 2022 Jun 14. PMID 35699578
- [Derived] Swift AJ, Wilson F, Cogliano M, Kendall L, Alandejani F, Alabed S, Hughes P, Shahin Y, Saunders L, Oram C, Capener D, Rothman A, Garg P, Johns C, Austin M, Macdonald A, Pickworth J, Hickey P, Condliffe R, Cahn A, Lawrie A, Wild JM, Kiely DG. Repeatability and sensitivity to change of non-invasive end points in PAH: the RESPIRE study. Thorax. 2021 Oct;76(10):1032-1035. doi: 10.1136/thoraxjnl-2020-216078. Epub 2021 Feb 25. PMID 33632769